CLINICAL TRIAL: NCT04304521
Title: Fluid Responsiveness Predicted by a Stepwise PEEP Elevation Recruitment Maneuver in Mechanically Ventilated Patients, a Pilot Study
Brief Title: Fluid Responsiveness Predicted by a Stepwise PEEP Elevation Recruitment Maneuver in Mechanically Ventilated Patients
Acronym: STEP-PEEP
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN902018/CHUSTE
Record Dates: First submitted 2020-03-09; First posted 2020-03-11 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Mechanical Ventilation; Respiration, Artificial
Keywords: Mechanical Ventilation; Lung recruitment maneuver; central venous pressure; pulse pressure; stroke volume; fluid responsiveness
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intensive care: Patients admitted in the intensive care unit of the University Hospital of Saint-Etienne, France between December 2018 and July 2019
  Interventions: Procedure: Lung recruitment maneuver

INTERVENTIONS:
Procedure: Lung recruitment maneuver — Lung recruitment maneuver is used to reopen or prevent collapsed lung under mechanical ventilation so as to decrease respiratory complications. LRM induces a transient increase in intra-thoracic pressure and decreases in venous return, leading to a decrease in left ventricular end-diastolic area and stroke volume.

SUMMARY:
Hemodynamic and fluid optimization during perioperative period can reduce postoperative morbidity. The assessment of preload and determination of whether the patient is fluid responsive is still challenging. Static preload indices such as central venous pressure are not accurate to assess fluid responsiveness contrary to dynamic preload indices such as pulse pressure variation (PPV) and stroke volume (SV) variation. However, such indices suffer from several limitations and should be used under strict conditions. Alternative dynamic methods such as lung recruitment maneuvers (LRM) have been developed LRM can be used to reopen or prevent collapsed lung under mechanical ventilation so as to decrease respiratory complications. LRM induces a transient increase in intra-thoracic pressure and decreases in venous return, leading to a decrease in left ventricular end-diastolic area and stroke volume. Several studies have shown that the PEEP-induced decrease in stroke volume is related to pre-existing preload responsiveness. Few studies have also shown that LRM can represent a functional test to predict fluid responsiveness. However, monitoring stroke volume during LRM to assess fluid responsiveness is costly, and cardiac output devices may not be reliable. In this context, central venous pressure (CVP) or systemic arterial parameters monitoring are easily accessible and inexpensive during major surgery.

DETAILED DESCRIPTION:
The aims of the current study were

1. to assess the ability of a LRM with a stepwise increase of PEEP to predict fluid responsiveness in mechanically ventilated patients,
2. to identify the best criteria for fluid responsiveness prediction between variations of systolic aortic pressure (SAP), mean arterial pressure (MAP), diastolic aortic pressure (DAP), pulse pressure (PP) and central venous pressure (CVP),
3. to compare the ability of these criteria with pulse pressure variation (PPV) to predict fluid responsiveness

ELIGIBILITY:
Inclusion Criteria:

* needing invasive arterial blood pressure and pulse contour analysis (PICCO system) for cardiac output measurement,
* central venous pressure monitoring,
* using of protective mechanical ventilation
* Indication for fluid expansion
* Admitted in the intensive care unit of CHU of St ETienne

Exclusion Criteria:

* right ventricular dysfunction
* significant valvulopathy,
* ejection fraction less than 50%,
* arrhythmia
* contraindication to LRMs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admited in the intensive care unit of the University Hospital of Saint-Etienne
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
pulse pressure (mmHg) | At the inclusion
  Pulse pressure = systolic aortic pressure - diastolic aortic pressure
systolic aortic pressure (mmHg) | At the inclusion
diastolic aortic pressure (mmHg) | At the inclusion

SECONDARY OUTCOMES:
mean arterial pressure (mmHg) | At the inclusion
Stroke volume (ml) | At the inclusion
central venous pressure (mmHg) | At the inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain VALLIER, PhD, Principal Investigator — CHU de St Etienne
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vallier S, Bouchet JB, Desebbe O, Francou C, Raphael D, Tardy B, Gergele L, Morel J. Slope analysis for the prediction of fluid responsiveness by a stepwise PEEP elevation recruitment maneuver in mechanically ventilated patients. BMC Anesthesiol. 2022 Jan 3;22(1):4. doi: 10.1186/s12871-021-01544-x. PMID 34979928